CLINICAL TRIAL: NCT06570265
Title: Evaluation of Resorption, Safety, and Efficacy of Absorbable Collagen Membrane in Preventing Significant Bone Loss Following GBR (Guided Bone Regeneration) Procedure.
Brief Title: RES-SAFE (Resorption, Safety, and Efficacy of Absorbable Collagen Membrane)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hyundai Bioland Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC-MD-CIP-001
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Guided Bone Regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental)
  Interventions: Device: GBR membrane

INTERVENTIONS:
Device: GBR membrane — GBR procedure is a technique often used in conjunction with dental implants to enhance the success and stability of the implant. This technique involves using barrier membranes to protect the bone graft or defect site from the rapid proliferation of surrounding soft tissues. In this clinical investigation resorbable, collagen membrane will be used.

SUMMARY:
The clinical study aims to assess the long-term safety and efficacy of the interventional medical device. The clinical study will enrol up to 50 patients aged 18 years and older, who meet specific inclusion and exclusion criteria designed to ensure patient safety and reliable data collection.

ELIGIBILITY:
Inclusion Criteria (among others):

* Patients over 18 years old (both sex) with full legal capacity who understand the treatment and sign the informed consent and who are medically healthy, except treated condition.

Exclusion Criteria (among others):

* Patients with dental diseases or conditions (except treated condition);
* Patients with unsatisfactory oral hygiene;
* Patients with alcohol, substance abuse, smoking habits, known allergy to collagen;
* Patients with severe or chronic diseases or with systemic inflammation and all patients classified as unhealthy;
* Pregnant or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2026-05-16 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of collagen membrane's - efficacy and safety. | 6 months after intervention
  Remnants of the collagen membrane, new blood vessels formation, and the absence of inflammation in histological results.

SECONDARY OUTCOMES:
Complication rate | 7 days and 6 months after intervention
  Complication rate assessed as the ratio patients with any complication to all patients.
Change in bone dimensions | Baseline, 6 and 12 months after intervention
  % change in horizontal bone dimensions at three subcrestal levels assessed via CBCT.
VAS scale | On the day of intervention and after 1, 2, 3 days. Satisfaction - on the day of intervention.
  Scale VAS for pain, swelling, bleeding. VAS scale will be used to assess satisfaction of the intervention.
Assessment of collagen membrane's - safety. | From the beginning till the end.
  Number of (S)AEs.